CLINICAL TRIAL: NCT02971410
Title: Overcoming Chemotherapy Resistance in Refractory Multiple Myeloma With Simvastatin, A Pilot Study
Brief Title: Simvastatin in Overcoming Chemotherapy Resistance in Patients With Relapsed or Refractory Multiple Myeloma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI no longer interested in pursuing study.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00040660; NCI-2016-01465 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 26216 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-11-23 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Simvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (simvastatin) (Experimental): Patients receive standard of care chemotherapy for up to 3 courses and simvastatin (PO) daily 2 days before the first dose of chemotherapy for up to 2 days after the last dose of chemotherapy. Treatment with simvastatin continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Simvastatin

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Simvastatin — Given PO
  Other Names: MK 733; Synvinolin; Zocor

SUMMARY:
This pilot clinical trial studies how well simvastatin works in overcoming chemotherapy resistance in patients with multiple myeloma that has come back or does not respond to treatment. Simvastatin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the effect of simvastatin on myeloma (M)-protein and/or free light chains ratio when added to conventional chemotherapy for the treatment of multiple myeloma patients who have received up to 3 (=< 3) and > 3 different chemotherapy regimens. (group A and group B)

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS), time to progression (TTP), and duration of response (DOR) in group A, group B, and both groups combined.

II. To describe toxicities (frequency and severity during the treatment) in group A, group B, and both groups combined.

III. To estimate overall response (OR) in group A, group B, and both groups combined.

IV. To evaluate the quality of life (QoL) of patients on the combined treatment in group A, group B, and both groups combined.

OUTLINE:

Patients receive standard of care chemotherapy for up to 3 courses and simvastatin orally (PO) daily 2 days before the first dose of chemotherapy for up to 2 days after the last dose of chemotherapy. Treatment with simvastatin continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3-5 weeks for the first 6 months, and every 1-3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a definitive diagnosis of multiple myeloma (using the International Myeloma Working Group Guidelines)
* Patients must meet one of the following two requirements:

  * Have achieved minimal response (MR) or stable disease (SD) in current treatment regimen after receiving a minimum of two cycles
  * Have a partial response but show a decrease less than 25% or an increase less than 25% in measurable disease over a two month period

    * NOTE: Patients may be refractory to primary therapy or relapsed and have measurable or assessable disease; (refractory disease is defined as anything less than partial response [PR] or progression within 60 days of completing therapy)
* Patients with multiple myeloma must have measurable disease; measurable disease may be paraprotein in serum or urine or the presence of free light chains in serum or urine defined by one or more of the following criteria:

  * Presence of serum M-protein concentration > 1 g/dL
  * Urine M-protein excretion > 200 mg in 24-hour urine collection
  * Serum free light chain concentration >= 10 mg/dL and abnormal kappa/lambda ratio
  * Urine free light chain concentration >= 100 mg/L and abnormal kappa/lambda ratio
* If female patient with reproductive capacity: on effective means of barrier birth control during the entire duration of the treatment
* Eastern Cooperative Oncology Group (ECOG) or Karnofsky performance status of 0, 1, or 2 (Karnofsky >= 60%)
* Life expectancy of greater than 8 weeks
* Absolute neutrophil count >= 500/ul
* Platelets >= 30,000/ul
* Total bilirubin < 2 times the upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) < 3 x upper limit of normal
* Patients must have adequate renal function as defined by a creatinine clearance >= 40 mL/min (measured or estimated by the Cockcroft-Gault formula)
* Patients must have no signs of significant rhabdomyolysis determined by creatine phosphokinase (CPK) levels with a creatine kinase (CK) < 5 times the upper limit of normal
* Patients must have recovered from acute toxicities resulting from therapy administered prior to entering this study to grade 1 or less (Common Terminology Criteria for Adverse Events [CTCAE] 4); alopecia may be unresolved
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Patients who have not received any chemotherapy treatment for multiple myeloma prior to being enrolled in the study
* Patients who have no measureable disease by serologic or urine markers (detectable disease only by bone marrow or imaging scans)
* Patients who show progressive disease or are not tolerating the current chemotherapy regimen
* Patients who were receiving simvastatin (dose > 40 mg/day) while receiving current chemotherapy regimen for multiple myeloma
* Patients receiving any other investigational agent(s)
* Active second malignancy in the last 3 years except for non-melanoma skin cancer or carcinoma-in-situ
* History of hypersensitivity reactions attributed to simvastatin
* Patients receiving medications that may increase risk of rhabdomyolysis such as itraconazole, ketoconazole, erythromycin, cyclosporine, amiodarone, verapamil, clarithromycin, nefazodone, ranolazine, human immunodeficiency virus (HIV) protease inhibitors, gemfibrozil, posaconazole, danazol, amiodarone, diltiazem, and amlodipine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myopathy, untreated hypothyroidism, hereditary myopathy in the family history, unstable angina pectoris, liver disease not due to multiple myeloma, cardiac arrhythmia that is symptomatic or not rate controlled, active connective tissue disease, active autoimmune disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are ineligible, as treatment involves unforeseeable risks to the embryo or fetus; female patients with reproductive capacity are required to use effective means of birth control during the entire duration of the treatment
* Patients who have been on a statin other than simvastatin within 2 weeks of starting treatment on current study; these include atorvastatin, fluvastatin, lovastatin, pitavastatin, pravastatin, and rosuvastatin; if patient is on statin, will need to stop treatment 2 weeks prior to starting treatment on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in free light chain ratios | Up to 126 Days
  The success rate will be estimated overall and within the strata groups and 95% confidence intervals will be calculated around the estimate. Will also estimate the change in free light chain ratios and provide confidence intervals for those estimates, both overall and within groups.
Change in M-protein level measured using electrophoresis | Up to 126 Days
  The success rate will be estimated overall and within the strata groups and 95% confidence intervals will be calculated around the estimate. Will also estimate the change in M-proteins and provide confidence intervals for those estimates, both overall and within groups.

SECONDARY OUTCOMES:
DOR | Up to 28 months
  Will estimate the mean duration of response and provide confidence intervals in the subset of patients who respond. The proportion (with confidence interval) of subjects achieving a clinical benefit response will be calculated.
Incidence of toxicities evaluated according to National Cancer Institute CTCAE version 4.0 | Up to 28 months
  Toxicity data (both frequency and severity) will be summarized descriptively by showing the number of subjects experiencing each type of toxicity by grade for those with a grade 2 or higher.
OR including stringent complete remission (CR), CR, Partial Remission (PR), and very good PR | Up to 28 months
  The proportion (with confidence interval) of subjects achieving a clinical benefit response will be calculated.
Overall survival | Up to 28 months
  Will be analyzed initially using Kaplan-Meier estimation.
PFS | Up to 28 months
  Will be analyzed initially using Kaplan-Meier estimation.
QoL assessed using a survey designed by European Organization for Research and Treatment of Cancer (EORTC) | Up to 126 Days
  Quality of life outcomes from the EORTC survey will be summarized descriptively.
Response in patients who did and did not receive zoledronic acid with therapy | Up to 28 months
  Subset analysis will be done on patients who received zoledronic acid as part of their treatment while on study vs those who did not receive zoledronic acid to assess differences in response.
Time to first response | Up to 28 months
  Will be analyzed initially using Kaplan-Meier estimation.
Time to next therapy | Up to 28 months
  Will be analyzed initially using Kaplan-Meier estimation.
TTP | Up to 28 months
  Will be analyzed initially using Kaplan-Meier estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Rodriguez, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States